CLINICAL TRIAL: NCT02659098
Title: A Phase 2b, Multicenter, Double-masked, Randomized Study Evaluating the Safety and Clinical Response of Subretinal Administration of CNTO 2476 in Subjects With Visual Acuity Impairment Associated With Geographic Atrophy Secondary to Age Related Macular Degeneration
Brief Title: A Study to Evaluate the Safety and Clinical Response of Subretinal Administration of CNTO 2476 in Participants With Geographic Atrophy
Acronym: PRELUDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR106814; CNTO2476MDG2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-12-07; First posted 2016-01-20 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Visual Acuity; Geographic Atrophy; Macular Degeneration
Keywords: Best Corrected Visual Acuity; Geographic Atrophy; Macular Degeneration; CNTO 2476
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label Safety Run-in Phase: Treatment Group (Experimental): Participants will receive CNTO 2476 3.0 x 10^5 cells in 50 microliter (mcL). CNTO 2476 will be delivered using the custom-designed Delivery System.
  Interventions: Drug: CNTO 2476 3.0 x 10^5 cells; Device: Subretinal Delivery System

INTERVENTIONS:
Drug: CNTO 2476 3.0 x 10^5 cells — Participants will receive a single subretinal administration of CNTO 2476 3.0 x 10^5 cells in 50 microliter (mcL) given by subretinal Delivery System.
Device: Subretinal Delivery System — Participants will receive CNTO 2476 by using the Delivery System.

SUMMARY:
The purpose of this study is to evaluate the safety and performance profile of the suprachoroidal surgical approach and the Delivery System.

DETAILED DESCRIPTION:
This is a multicenter (when more than one hospital or medical school team work on a medical research study) study which includes an initial unmasked safety phase. The duration of participation in the study for each participant is approximately 3 years. Efficacy will be evaluated at 6 months, 12 months and annually thereafter. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of geographic atrophy (GA) secondary to age-related macular degeneration (AMD) confirmed within 45 days prior to initial randomization verified by the central reading center
* Study eyes will have a best corrected visual acuity (BCVA) of 20/80 to 20/800 [Early Treatment Diabetic Retinopathy Study (ETDRS) log of the minimum angle of resolution (logMAR) value 0.6-1.6]. The treatment eye will be that with the worse BCVA at Screening. If BCVA is clinically equivalent, the eye with the larger GA determines the study eye
* Participant is a suitable candidate for ophthalmologic surgery, is willing and able to comply with the surgical procedure, scheduled visits, treatment plan, laboratory tests and other study procedures. Participant has met criteria of the surgery center anti-coagulation protocol, if applicable
* Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Participant has a history of neovascular ("wet") AMD in the treatment eye, including evidence of retinal pigment epithelium rips or evidence of subretinal or choroidal neovascularization or fluid. In cases where imaging is inconclusive, review of the case with the study site, considering history and imaging will determine eligibility. History or evidence of neovascular AMD in the fellow eye is allowed, if anti-vascular endothelial growth factor (VEGF) therapy has not been required for at least 8 weeks prior to Screening
* Geographic atrophy secondary to any causes other than AMD in either eye
* A diagnosis of glaucoma with an intraocular pressure (IOP) greater than or equal to (>=) 25 millimeter of mercury (mmHg) while being treated with an ocular hypotensive drug. Treatment should be no more than 1 drug preparation/combination, which can contain 1 or 2 ocular hypotensive active ingredients; participants receiving more than 2 ocular hypotensive active ingredients are excluded
* Nuclear sclerotic cataract, cortical spoking, posterior subcapsular cataract above Grade 2 per Age Related Eye Disease Study (AREDS) scale or any other ophthalmologic condition that reduces the clarity of the media that, in the opinion of the investigator or reading center, interferes with ophthalmologic examination (example, corneal abnormalities, inadequate pupillary dilation), surgery or imaging in the study eye
* Myopia greater than minus (>-) 8 diopters and participants with greater than (>) 4 diopters of astigmatism, and greater than plus (>+) 10 diopters of hyperopia

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- United States (8):
  - Arcadia, California
  - Chicago, Illinois
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Royal Oak, Michigan
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- CNTO 2476 3.0*10^5 Cells: Participants received a single subretinal administration of CNTO 2476 (Palucorcel) comprising 3.0*10^5 cells in 50 microliters (mcL) dosing volume on Day 1. CNTO 2476 was delivered using the custom-designed Delivery System and surgical procedure.
Period: Overall Study
Arm/Group | CNTO 2476 3.0*10^5 Cells
Started | 21
Completed | 14
Not Completed | 7
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.9 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Total Letters Score at Month 1- Treated Eye
Description: Best corrected visual acuity (BCVA) was assessed in the study eye (Treated eye). BCVA measurements were made using the logarithm of the minimum angle of resolution (logMAR) visual acuity testing charts. Each letter on the chart has a score value of 0.02 log units. Since there were 5 letters per line, the total score for a line on the logMAR chart represented a change of 0.1 log units. The formula for calculating the logMAR BCVA score was: 1.7 - 0.02*number of letters read. A lower BCVA score indicates better vision. A negative change score indicates improvement.
Time Frame: Baseline and Month 1
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
logMAR | 0.132 (0.2093)

2. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 2- Treated Eye
Description: BCVA was assessed in the study eye (Treated eye). BCVA measurements were made using the logMAR visual acuity testing charts. Each letter on the chart has a score value of 0.02 log units. Since there were 5 letters per line, the total score for a line on the logMAR chart represented a change of 0.1 log units. The formula for calculating the logMAR BCVA score was: 1.7 - 0.02*number of letters read. A lower BCVA score indicates better vision. A negative change score indicates improvement.
Time Frame: Baseline and Month 2
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
logMAR | 0.073 (0.2273)

3. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 3- Treated Eye
Description: as for outcome 2
Time Frame: Baseline and Month 3
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
logMAR | 0.079 (0.2502)

4. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 6- Treated Eye
Description: as for outcome 2
Time Frame: Baseline and Month 6
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
logMAR | 0.090 (0.2628)

5. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 12- Treated Eye
Description: as for outcome 2
Time Frame: Baseline and Month 12
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study. Here, N (number of participants analyzed) signifies number of participant evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 18
logMAR | 0.119 (0.2598)

6. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 18- Treated Eye
Description: as for outcome 2
Time Frame: Baseline and Month 18
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 17
logMAR | 0.107 (0.2512)

7. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Total Letters Score at Month 24- Treated Eye
Description: as for outcome 2
Time Frame: Baseline and Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 15
logMAR | 0.145 (0.3065)

8. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Total Letters Score at Month 30- Treated Eye
Description: as for outcome 2
Time Frame: Baseline and Month 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 13
logMAR | 0.112 (0.3093)

9. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Total Letters Score at Month 36- Treated Eye
Description: as for outcome 2
Time Frame: Baseline and Month 36
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 13
logMAR | 0.211 (0.3639)

10. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Total Letters Score at Month 1- Fellow Eye
Description: BCVA was assessed in the fellow eye. BCVA measurements were made using the logMAR visual acuity testing charts. Each letter on the chart has a score value of 0.02 log units. Since there were 5 letters per line, the total score for a line on the logMAR chart represented a change of 0.1 log units. The formula for calculating the logMAR BCVA score was: 1.7 - 0.02*number of letters read. A lower BCVA score indicates better vision. A negative change score indicates improvement.
Time Frame: Baseline and Month 1
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
logMAR | 0.017 (0.0962)

11. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 2- Fellow Eye
Description: as for outcome 10
Time Frame: Baseline and Month 2
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
logMAR | 0.027 (0.0868)

12. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 3- Fellow Eye
Description: as for outcome 10
Time Frame: Baseline and Month 3
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
logMAR | 0.010 (0.0960)

13. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 6- Fellow Eye
Description: as for outcome 10
Time Frame: Baseline and Month 6
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
logMAR | 0.033 (0.1351)

14. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 12- Fellow Eye
Description: BCVA was assessed in the fellow eye. BCVA measurements were made using logMAR visual acuity testing charts. Each letter on the chart has a score value of 0.02 log units. Since there are 5 letters per line, the total score for a line on the logMAR chart represents a change of 0.1 log units. The formula for calculating the logMAR BCVA score is: 1.7 - 0.02*number of letters read. A lower BCVA score indicates better vision. A negative change score indicates improvement.
Time Frame: Baseline and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 18
logMAR | 0.074 (0.1807)

15. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 18- Fellow Eye
Description: as for outcome 10
Time Frame: Baseline and Month 18
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 17
logMAR | 0.075 (0.1728)

16. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 24- Fellow Eye
Description: as for outcome 10
Time Frame: Baseline and Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 15
logMAR | 0.115 (0.1962)

17. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 30- Fellow Eye
Description: as for outcome 10
Time Frame: Baseline and Month 30
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 14
logMAR | 0.106 (0.1721)

18. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity Total Letters Score at Month 36- Fellow Eye
Description: as for outcome 10
Time Frame: Baseline and Month 36
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 13
logMAR | 0.309 (0.2435)

19. Secondary Outcome: Percentage of Participants Losing Greater Than or Equal to (>=) 15 Best Corrected Visual Acuity Letters: Treated Eye
Description: BCVA was assessed as letters read using early treatment diabetic retinopathy study charts and reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye (Treated eye). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. The percentage of participants losing >=15 BCVA in the study eye were reported.
Time Frame: Months 1, 2 , 3, 6, 12, 18, 24, 30 and 36
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study. Here 'n' (number analyzed) signifies the number of participants who had BCVA data at a visit.
Measure: Number; unit: Percentage of Participants
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
Percentage of Participants
  Month 1: Week 4 | 14.3
  Month 2 | 14.3
  Month 3 | 19.0
  Month 6 | 14.3
  Month 12: number analyzed (Participants) | 18
  Month 12 | 16.7
  Month 18: number analyzed (Participants) | 17
  Month 18 | 17.6
  Month 24: number analyzed (Participants) | 15
  Month 24 | 20.0
  Month 30: number analyzed (Participants) | 13
  Month 30 | 23.1
  Month 36: number analyzed (Participants) | 13
  Month 36 | 30.8

20. Secondary Outcome: Percentage of Participants Losing >=15 Best Corrected Visual Acuity Letters: Fellow Eye
Description: BCVA was assessed as letters read using early treatment diabetic retinopathy study charts and reported as the number of letters read correctly (ranging from 0 to 100 letters) in the fellow eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. The percentage of participants losing >=15 BCVA in the fellow eye were reported.
Time Frame: Months 1, 2 , 3, 6, 12, 18, 24, 30 and 36
Population: as for outcome 19
Measure: Number; unit: Percentage of Participants
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
Percentage of Participants
  Month 1: Week 4 | 0
  Month 2 | 0
  Month 3 | 0
  Month 6 | 4.8
  Month 12: number analyzed (Participants) | 18
  Month 12 | 16.7
  Month 18: number analyzed (Participants) | 17
  Month 18 | 17.6
  Month 24: number analyzed (Participants) | 15
  Month 24 | 13.3
  Month 30: number analyzed (Participants) | 14
  Month 30 | 14.3
  Month 36: number analyzed (Participants) | 13
  Month 36 | 46.2

21. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity Letters at Months 6 and 12: Treated Eye
Description: BCVA was assessed as letters read using early treatment diabetic retinopathy study charts and reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye (Treated eye). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening.
Time Frame: Baseline, Months 6 and 12
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study. Here 'n' (number analyzed) signifies the number of participants analyzed at the specified time point.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
Letters
  Month 6 | -4.5 (13.14)
  Month 12: number analyzed (Participants) | 18
  Month 12 | -5.9 (12.99)

22. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity at Months 6 and 12: Fellow Eye
Description: BCVA was assessed as letters read using early treatment diabetic retinopathy study charts and reported as the number of letters read correctly (ranging from 0 to 100 letters) in the fellow eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening.
Time Frame: Baseline, Months 6 and 12
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
Letters
  Month 6 | -1.7 (6.76)
  Month 12: number analyzed (Participants) | 18
  Month 12 | 6.76 (9.03)

23. Secondary Outcome: Change From Baseline in Growth Rate of Geographic Atrophy (GA) Lesion Area at Months 6 and 12: Treated Eye
Description: The area of GA was determined based primarily on fundus autofluorescence (FAF). The change in GA lesion area was measured by FAF and analysis of FAF images was performed by the central reading center. A positive change from baseline indicates an increase in size of GA lesion area (worsening; disease progression).
Time Frame: Baseline, Months 6 and 12
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study. Here, N (number of participants analyzed) signifies number of participant evaluable for this endpoint and 'n' (number analyzed) signifies the number of participants analyzed at the specified time point.
Measure: Mean (Standard Deviation); unit: Square millimeter
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 17
Square millimeter
  Month 6 | 0.6691 (2.3301)
  Month 12: number analyzed (Participants) | 11
  Month 12 | 2.4214 (1.3661)

24. Secondary Outcome: Change From Baseline in Growth Rate of Geographic Atrophy Lesion Area at Months 6 and 12: Fellow Eye
Description: The area of GA was determined based primarily on FAF. The change in GA lesion area was measured by FAF and analysis of FAF images was performed by the central reading center. A positive change from baseline indicates an increase in size of GA lesion area (worsening; disease progression).
Time Frame: Baseline, Months 6 and 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Square millimeter
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 13
Square millimeter
  Month 6: number analyzed (Participants) | 12
  Month 6 | 1.2085 (0.7060)
  Month 12 | 2.6457 (1.9449)

25. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Number of participants with TEAEs and SAEs were assessed. An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment and can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product. SAE is defined as any untoward medical occurrence that at any dose results in death, Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent or significant disability/incapacity, Is a congenital anomaly/birth defect, Is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Up to Months 36
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
Participants
  Treatment-emergent Adverse Events | 20
  Treatment-emergent Serious Adverse Events | 5

26. Secondary Outcome: Number of Participants With Ocular Treatment-emergent Adverse Events
Description: Number of participants with ocular TEAE were assessed. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment and can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product.
Time Frame: Up to Months 36
Population: The safety analysis set defined as participants who were enrolled and received surgery in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | CNTO 2476 3.0*10^5 Cells
Number analyzed (Participants) | 21
Participants
  Treated Eye | 17
  Fellow Eye | 10

ADVERSE EVENTS:
Time Frame: Up to 36 Months
Description: The safety analysis set defined as participants who were enrolled and received surgery in the study.
Arm/Group | CNTO 2476 3.0*10^5 Cells
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CNTO 2476 3.0*10^5 Cells (N=21)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1
Aortic Valve Stenosis (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CNTO 2476 3.0*10^5 Cells (N=21)
Atrial Fibrillation (Cardiac disorders) | 2
Anterior Chamber Cell (Eye disorders) | 2
Cataract (Eye disorders) | 2
Cataract Nuclear (Eye disorders) | 3
Charles Bonnet Syndrome (Eye disorders) | 2
Conjunctival Haemorrhage (Eye disorders) | 9
Conjunctival Oedema (Eye disorders) | 2
Neovascular Age-Related Macular Degeneration (Eye disorders) | 3
Retinal Haemorrhage (Eye disorders) | 7
Visual Acuity Reduced (Eye disorders) | 5
Visual Impairment (Eye disorders) | 2
Vitreous Detachment (Eye disorders) | 2
Vitreous Floaters (Eye disorders) | 4
Sensation of Foreign Body (General disorders) | 5
Urinary Tract Infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Corneal Abrasion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Hypertension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Protocol Amendment 3 eliminated 2nd safety cohort and randomized masked portion of study per Sponsor decision to terminate development. Protocol specified follow-up visits were completed for treated participants, thus study was considered completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT02659098/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT02659098/SAP_001.pdf